CLINICAL TRIAL: NCT06594822
Title: Effectiveness of Probiotics and Standard Therapy Versus Standard Therapy Alone in Patients of Mild to Moderate Rheumatoid Arthritis
Brief Title: Effectiveness of Probiotics in Patients of Mild to Moderate Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fawad Ahmad Randhawa, Associate Professor of Endocrinology, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8864/KEMU/2023
Record Dates: First submitted 2024-08-18; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
Keywords: DAS-28; Probiotics; EULAR; NSAIDs; DMARDs; RF; anti-CCP; hsCRP; CBC; LFTs; RFTs; SPSS
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Probiotics; Anti-Inflammatory Agents, Non-Steroidal; Glucocorticoids; Antirheumatic Agents

STUDY DESIGN:
Intervention Model Description: Simple random selection of patients. Assigned to 2 groups by computer generated method. Group A received standard treatment of analgesics, glucocorticoids and methotrexate and or sulfasalazine. Group B was the interventional group that received probiotics in addition to standard treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A, Probiotic Group (Experimental): Probiotics were given as an adjunct to standard therapy i.e., NSAIDs, Steroids, DMARDs
  Interventions: Dietary Supplement: probiotic plus standard treatment
- Group B, Standard treatment group (Active Comparator): Standard therapy including NSAIDs, steroids and DMARDs
  Interventions: Drug: standard treatment

INTERVENTIONS:
Dietary Supplement: probiotic plus standard treatment — Bacillus clausii, 5ml ampule containing 2 billion spores, given orally once daily
  Arms: Group A, Probiotic Group
Drug: standard treatment — diclofenac 50 mg twice a day, prednisone 5mg once daily, methotrexate 10mg once weekly or sulfasalazine 500 twice daily
  Other Names: NSAID, glucocorticoid and DMARD
  Arms: Group B, Standard treatment group

SUMMARY:
To assess the effectiveness of probiotics when given in combination with standard therapy in patients of mild to moderate rheumatoid arthritis

DETAILED DESCRIPTION:
This study was conducted on the patients presenting to the Rheumatology out-patients department of the Department of Medicine, King Edward Medical University, Mayo hospital, Lahore from 24th August, 2023 till 23rd February, 2024. A total of 88 patients of either sex, between the age group of 18 to 70 years and having an established diagnosis of rheumatoid arthritis (RA), [as proved on history, X-rays and biologic markers like Rheumatoid Factor (RF) and Anti-cyclic citrullinated protein antibodies (anti-CCP antibodies), Erythrocyte Sedimentation Rate (ESR) and C- reactive protein (CRP)] and having mild to moderate disease activity score (DAS-28 score between 2.6 to <5.1) were selected via simple random sampling.

After approval from the Board of Studies (BOS) and Advanced Study Research Board (ASRB) of King Edward Medical University, Mayo Hospital, Lahore, all patients conforming to the selection criteria were enrolled in the study. Informed written and verbal consent was taken from all the participants. Patient's demographic data was obtained and recorded in a predesigned proforma. Patients were divided into two groups by computer generated method. Group A comprised 44 patients who received standard therapy [analgesics, glucocorticoids, any Disease modifying anti-rheumatic drug (DMARD)] alongwith probiotic (Bacillus clausii), whereas Group B also comprising 44 patients received standard therapy alone. Lab investigations like complete blood counts (CBC), C- reactive protein (CRP), liver function tests (LFTs) and renal function tests (RFTs) were done at baseline and then on follow up visits at 45 and 90 days. Disease activity score (DAS-28) was assessed on baseline then on each subsequent visit to monitor response to treatment. Mild RA patients had a DAS-28 score between 2.6 to 3.1 and moderate RA patients had a DAS-28 score between 3.1 to <5.1. Effectiveness was defined in terms of reduction of DAS-28 score of ≥0.6 from the baseline based on European League against Rheumatism (EULAR) response rates. Pancytopenia, derangement in LFTs and RFTs twice from the baseline as a result of treatment resulted in exclusion from the study.

Data was analyzed using computer software Statistical Package for Social Sciences (SPSS) version 26.0. Quantitative variables like age, DAS-28 score were expressed as mean and standard deviation (Mean±SD). Qualitative variables including gender were expressed as frequency and percentages. Chi- square test was used to compare response between the two groups. P value ≤0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: 1- Patients of either sex. 2- Patients between the age group of 18 to 70 years. 3- Patients having an established diagnosis of rheumatoid arthritis (proven on history, X-rays and biologic markers like RF and Anti-CCP antibodies, ESR and CRP).

4- Patients having mild to moderate disease activity (DAS-28 score between 2.6 to <5.1).

Exclusion Criteria:1- Patients treated previously for RA with probiotics. 2- Patients with a history of allergy to probiotics. 3- Patients with mixed connective tissue disorder and overlap syndrome as per history and labs.

4- Patients with a history of gastrectomy, renal failure and liver cirrhosis. 5- Patients with recent or current use of antibiotics. 6- Pregnant patients and lactating mothers.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score (DAS-28) score | 3 months
  Reduction in DAS-28 score of ≥ 0.6 from the baseline. (Mild RA baseline score between 2.6 - 3.1, Moderate RA baseline score between 3.1 to <5.1)

CONTACTS AND LOCATIONS:
Overall Officials: Gulraiz Iqbal, MBBS, Principal Investigator — King Edward Medical University
Locations (1):
- Tazeen Nazar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No